CLINICAL TRIAL: NCT05906147
Title: Health ImprOvement Program of Bone in China
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, sheng zhifeng, Director of the Health Management Center of the Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Other Study IDs: LYF2021015.
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Regular follow-up — Follow-up of the population was conducted to track the incidence of fractures

SUMMARY:
Fracture risk factors have long been identified as key factors in osteoporosis and fragility fractures. The WHO recommended Fracture risk assessmenttool (FRAX) applies clinical risk factors to assess the absolute risk of osteoporotic fractures in each individual. Our preliminary study suggests that FRAX estimates may underestimate the risk of fractures in the Chinese population. In order to optimize the risk prediction model of osteoporotic fractures, a treatment threshold and its optimal cutting point were initially established based on the data of the health management Center of the Second Xiangya Hospital of Central South University.

ELIGIBILITY:
Inclusion Criteria:

* Dual-energy X-ray bone mineral density measurement was performed in the health management center of our hospital in the physical examination subjects over 40 years old. Have independent civil capacity and agree to participate, and sign informed consent

Exclusion Criteria:

* Under 40 years of age， Patients who had undergone hip replacement or lumbar surgery and could not perform dual-energy X-ray BMD testing; Patients who have been treated with effective anti-osteoporosis drugs or have a history of malignant tumors.

Ages: 40 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Dual-energy X-ray bone mineral density measurement was performed in the health management center of our hospital in the physical examination subjects over 40 years old
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2031-02-27 (Estimated)

PRIMARY OUTCOMES:
bone mineral density bone mineral density | From 2021 to 2031
  Bone mineral density (BMD) data measured by dual-energy X-ray absorptiometry were collected from patients over 40 years old
Occurrence of fracture | From 2021 to 2031
  Follow-up of the population was conducted to track the incidence of fractures
clinical risk factors of osteoporotic fracture | From 2021 to 2031
  The main clinical risk factors of osteoporotic fracture were collected

CONTACTS AND LOCATIONS:
Locations (1):
- Health Management Center, The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided